CLINICAL TRIAL: NCT04728945
Title: Prevention of Perioperative Pulmonary Complications by Lung Recruitment During Laparoscopic Surgery in Trendelenburg Head-down Position
Brief Title: Prevention of Perioperative Pulmonary Complications by Lung Recruitment During Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Toho University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Reclap study
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Perioperative Complication; Hypoxia
Keywords: perioperative pulmonary complications; lung recruitment; laparoscopic surgery
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lung recruitment (Experimental): Standard ventilatory management with lung recruitment every 30 minutes
  Interventions: Procedure: lung recruitment; Procedure: Standard ventilatory management
- control (Active Comparator): Standard ventilatory management
  Interventions: Procedure: Standard ventilatory management

INTERVENTIONS:
Procedure: lung recruitment — Automatic lung recruitment using the anesthetic machines (with PEEP 15 cmH2O for 30 seconds) will be performed every 30 minutes during laparoscopy.
  Arms: lung recruitment
Procedure: Standard ventilatory management — After tracheal intubation, standard ventilatory management (metered ventilation) should be performed with the following initial settings, and rescue should be performed when hypoxemia occurs, if necessary.
  [initial setting] PEEP 4cmH2O, FIO2 0.3 Ventilation rate: 6-8 ml/kg predicted body weight (PBW)

SUMMARY:
Perioperative pulmonary complications such as atelectasis, hypoxemia, and pneumonia after ventilatory management during general anesthesia have a negative impact on patient outcomes. The possibility of reducing perioperative pulmonary complications by lung recruitment, which uses positive pressure to prevent alveolar collapse, has been reported. Although laparoscopic surgery, which has been widely performed in recent years, can reduce the invasiveness of the operation, it is prone to alveolar collapse due to increased abdominal pressure and diaphragm elevation. The purpose of this study is to verify whether the lung recruitment during laparoscopic surgery in Trendelenburg head-down position prevents hypoxemia due to lung collapse.

DETAILED DESCRIPTION:
The multi-center RCT will enroll 80 patients who have laparoscopic surgery in Trendelenburg head-down position. Informed consent will be obtained for study subjects who meet the selection criteria, and the subjects will be enrolled in Electronic Data Capture and randomized into two groups. Patients will be admitted to the operating room for induction of anesthesia and tracheal intubation. In the control group, mechanical ventilation will be performed according to the initial settings and protocols. In the intervention group, after intubation, the ventilator will be initially set up, and the first pulmonary recruitment will be performed immediately after the start of the laparoscopy, followed by recruitment every 30 minutes until the end of the laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing low head laparoscopic surgery who are expected to be laparoscopic for more than 2 hours

Exclusion Criteria:

* Lateral or supine position
* BMI > 35
* One-second rate <70%, %VC <80%, obstructive, restrictive, with bra
* Cardiovascular disease (NYHA III or higher)
* Intracranial hypertensive disease
* Emergency surgery
* Pregnancy
* Glaucoma
* Patients judged unsuitable by the anesthesiologist in charge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia | During laparoscopy procedure
  SpO2 less than 95% or more than 2% decrease from baseline
Time to onset of hypoxia | During laparoscopy procedure
  Duration from the start of laparoscopic surgery to the onset of hypoxia

SECONDARY OUTCOMES:
Rate of decrease in SpO2 | During laparoscopy procedure
  Difference between baseline SpO2 and minimum SpO2 during laparoscopic surgery
Ventilator setting at the end of surgery | During surgery
  Ventilator settings such as FIO2, PEEP, and plateau pressure
compliance rate of lung recruitment | During laparoscopy procedure
  compliance rate of lung recruitment in the intevention group
Safety endpoint: Circulatory agonist use | During surgery
  Circulatory agonist use
Safety endpoint: total fluid infusion | During surgery
  total fluid infusion
Safety endpoint: incidence of complications | During surgery
  incidence of complications (hypotension, arrhythmia, pneumothorax, atelectasis defined by the blinded investigator)
Postoperative hypoxia | the day after surgery
  Presence of hypoxia the day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Fujino, Study Chair — Department of Anesthesiology and Intensive Care Medicine, Osaka University
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Osaka University, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No